CLINICAL TRIAL: NCT01804166
Title: A Research Study to Bank Samples for Future Evaluation to Identify Biomarkers That Predispose Crohn's Disease and Ulcerative Colitis Patients to Develop Hepatosplenic T-Cell Lymphoma (HSTCL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR100938; CR100938 (Registry Identifier: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2013-02-01; First posted 2013-03-05 (Estimated); Results first posted 2021-03-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Hepatosplenic T-Cell Lymphoma
Keywords: Lymphoma, T-Cell, Peripheral, Infliximab, Golimumab, Remicade, Simponi, Ulcerative Colitis, Crohn's Disease, Inflammatory Bowel Disease
MeSH Terms: conditions — Lymphoma; Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases | interventions — Infliximab; golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- IBD patients with HSTCL (Other): Subjects with Inflammatory Bowel Disease with a diagnosis of Hepatosplenic T-cell lymphoma
  Interventions: Drug: Infliximab; Drug: Golimumab

INTERVENTIONS:
Drug: Infliximab — This study will not restrict or introduce any therapeutic interventions, including medications. Participants may continue to receive infliximab as instructed by their personal physicians.
  Other Names: Remicade
Drug: Golimumab — This study will not restrict or introduce any therapeutic interventions, including medications. Participants may continue to receive golimumab as instructed by their personal physicians.
  Other Names: Simponi

SUMMARY:
This study is designed to collect tissue samples from the biopsy specimen that was used to diagnose hepatosplenic T-cell lymphoma (HSTCL), additional patient information, and if possible, to obtain additional samples including a single blood sample, a buccal swab sample and/or a bowel tissue sample. Samples obtained will be stored by the sponsor for future testing. In addition, demographic and clinical patient information will be collected. The study will be conducted in North America. Patients eligible for enrollment include males or females with IBD of any age who have a confirmed diagnosis of HSTCL. Patients will be identified through the sponsor's adverse event reporting systems. Cases reported to the sponsor's Medical Information Center will be queried to ascertain if the reporter is interested in participating in the study. Where appropriate, cases may also be identified through the sponsor's new or on-going clinical trials and registries. Samples may be collected from living patients or from stored tissue of deceased patients. This study will not restrict or introduce any therapeutic interventions, including medications. All patients will continue to be managed by their personal physicians. No healthy subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Inflammatory Bowel Disease with a confirmed diagnosis of Hepatosplenic T-cell Lymphoma
* Provide written informed consent (either by the patient or his/her legal representative). Consent from a legally acceptable representative of a deceased patient will be obtained for enrollment into the study and sample collection
* Be willing to provide a tumor biopsy sample for the study

Exclusion Criteria:

* Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (for example, compromise the well-being) of the patient or that could prevent, limit, or confound the protocol-specified assessments
* Is unable to provide critical clinical and/or demographic patient and/or sample information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-03-21 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Janssen Scientific Affairs, LLC
Locations (1):
- Norfolk, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 12 subjects the Sponsor attempted to enroll in the study, 1 subject consented and provided a biopsy sample for analysis. No subjects discontinued from the study after enrollment.
Period: Overall Study
Arm/Group | IBD Patients With HSTCL
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Since only one participant completed the study, due to confidentiality issues, no data will be reported.
Arm/Group | IBD Patients With HSTCL
Number analyzed (Participants) | 0
Age, Continuous [unit: Years]
Sex: Female, Male
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Number of Samples Collected for the Identification of Biomarkers for Early Evaluation of Risk of Developing Hepatosplenic T-cell Lymphoma (HSTCL)
Description: Samples will be collected from IBD patients diagnosed with HSTCL for future evaluation to identify biomarkers that may allow either earlier evaluation of a participant's risk of developing HSTCL or possibly earlier diagnosis.
Time Frame: Approximately up to 8 years
Population: Since only one participant completed the study, due to confidentiality issues, no data will be reported.
Arm/Group | IBD Patients With HSTCL
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately up to 8 years
Arm/Group | IBD Patients With HSTCL
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The low enrollment in this study combined with the limited published information related to biomarkers related to HSTCL limit the ability to interpret and apply any results from this study to the broader IBD population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (1):
  • Study Protocol (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT01804166/Prot_000.pdf